CLINICAL TRIAL: NCT03734185
Title: Cardiac Rehabilitation: From Hospital to Municipal Setting.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Defactum, Central Denmark Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: Cardiac Rehab
Record Dates: First submitted 2018-10-19; First posted 2018-11-07 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2022-06

CONDITIONS: Cardiac Rehabilitation
Keywords: Cardiac Rehabilitation
MeSH Terms: interventions — Educational Status; Coping Skills

STUDY DESIGN:
Masking Description: Included municipalities are expected to receive 2,310 patients with IHD per year (figures from 2017) to attend a CR program. Statistical power; These figures were used to address "the difference in patient outcome in intervention CR and usual CR". Using the minimally important difference available for HeartQoL (mean difference of 2.0, standard deviation 2.0)(1) and the HADS (mean difference of 2.0 and standard deviation of 3.8)(2) and within site clustering ( intra-cluster correlation of 0.01 and an average cluster size of 185 patients - design effect of 2.84) we would need to recruit at least 312 patients per group at 90% power and 5%.
  References
  1. Smid DE, et al. Responsiveness and MCID Estimates for CAT... J Am Med Dir Assoc 2017 Jan;18(1):53-58.
  2. Oldridge N, et al. The HeartQoL: Part II. Validation of a new core health-related quality of life questionnaire... Eur J Prev Cardiolog 2014 01/01; 2017/09;21(1):98-106.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Learning and Coping (Experimental): A health pedagogical strategy that builds on inductive teaching with high involvement of the participants. Characteristics of Learning and Coping are that 'experienced patients' plan, teach and evaluate, in cooperation with health professionals.
  Interventions: Other: Learning and Coping
- Usual Cardiac Rehabilitation (Active Comparator): The theoretical frameworks used in some of these local healthcare services are empowerment, self-efficacy and self-management
  Interventions: Other: Learning and Coping

INTERVENTIONS:
Other: Learning and Coping — 'Experienced patients' plan, teach and evaluate, in cooperation with health professionals.

SUMMARY:
In recent decades, local healthcare services have undergone dramatic changes. The World Health Organization (WHO) refers to a shift from specialized hospital to local healthcare services to meet the growing expectations for better performance and outcomes in health care and better value for money. It is unique that Central Denmark Region has assigned phase II cardiac rehabilitation (CR) as a local healthcare task. However, there is sparse knowledge about how this reform may influence processes of care and outcomes in CR. This association is important to investigate when dramatic organisational changes in settings of evidence based interventions is implemented, as well as in relation to helping people with heart disease return to an active and satisfying everyday life.

DETAILED DESCRIPTION:
Background In recent decades, local healthcare services have undergone dramatic changes. The World Health Organization (WHO) refers to a shift from specialized hospital to local healthcare services to meet the growing expectations for better performance and outcomes in health care and better value for money. In line with the WHO statements a structural reform reorganised the entire public sector in Denmark in 2007. The local healthcare services were given the responsibility for the more generalised rehabilitation of patients with chronic diseases, and hospitals were to carry out more specialised rehabilitation for patients with chronic diseases admitted to a hospital. Today, several local healthcare services provide non-pharmacological phase II cardiac rehabilitation (CR); this phase encompasses the immediate post discharged period. Central Denmark Region has - as the only region in Denmark - assigned phase II CR as a local healthcare task. This unique reform became effective on 1 January, 2017. However, there is sparse knowledge about how this reform may influence processes of care and outcomes in CR.

CR programmes do not meet the required evidence-based standard Several countries have developed clinical practice guidelines for CR, including Denmark in 2013. The guidelines incorporate the best available evidence for the management of CR to assist health professionals and patient decisions about appropriate rehabilitation. However, it is unclear to what extent local healthcare services CR is performed in accordance with the clinical practice guidelines for CR. Doherty P et al. studied the extent to which programmes meet national minimum standards for the delivery of CR as prescribed by the National Certification Programme for CR in UK. The authors found that 31% out of 170 unique CR programmes were delivered with high performance, 46% as mid-level performance, 18% were lower-level, while 5% failed to meet any of the minimum criteria. We have not been able to find other similar studies for performance of CR programmes in Denmark or elsewhere. Therefore, it is unclear whether the performance varies in local healthcare services CR programmes in Denmark, and whether there is a need for improvement to provide all patients a high-quality evidence-based service.

Patient education using learning and coping improves adherence Patient education is recommended in the clinical practice guidelines for CR and is defined as: "The process by which health professionals and others impact information to patients who will change their health behaviors or improve their health status". In the guidelines several educational topics are listed as important for patient education. However, the rationale for the specific areas is not completely explained in the guidelines. Furthermore, the guidelines only advice on what to teach, not how it should be done e.g. educational models, material, provider and setting. A systematic review shows that the delivery of patient education programmes can vary substantially, but common topics include nutrition, exercise, risk factor modification, psychosocial well-being and medications. Also duration, frequency and ongoing maintenance or re-inforcement vary between programmes. However, the Danish Health Authority recommend using evidence-based methods in patient education including Learning and Coping, Motivational interview.

In Central Denmark Region, six out of 19 local healthcare services have decided to use Learning and Coping in CR while remaining local healthcare services use different approaches. Learning and Coping is a health pedagogical strategy that builds on inductive teaching with high involvement of the participants. Characteristics of Learning and Coping are that 'experienced patients' plan, teach and evaluate, in cooperation with health professionals. In a hospital setting, Learning and Coping has shown an increase inpatient adherence in CR including training and patient education, especially for those with low socioeconomic status. However, it is unclear whether using Learning and Coping in local healthcare services performs similar results. These results are needed because low socioeconomic status is a common barrier to attending CR programmes.

Patient education using Learning and Coping to overcome barriers to CR System-, physical- and personal-level barriers in CR are well-described in the literature. Studies show that 13% to 20% of eligible patients are not referred to CR, and 19% to 45% do not attend CR. Also, long wait time to CR after referral entail low attendance. Health-related factors such as anxiety, depression, pain, or other illnesses are reported curtail the uptake. Like exercise-limiting comorbidities predict fewer sessions. Older adults, women, people who belong to ethnic minority groups, are young, have low socioeconomic status, live alone and receive limited social support are low attenders. Other studies show that family obligations and the distance from home to the programme setting entail low attendance. Few studies found that self-payment is a barrier to attend CR. This may not be an issue in Denmark as the Danish healthcare system provides tax-funded healthcare to the country's 5.7 million residents, including free access to hospital care, general practitioners and primary healthcare services including CR. Patients should be encouraged to attend patient education as literature reviews show that educational interventions with cardiac care increase patients' knowledge and facilitate behavior change. Furthermore, education interventions increase physical activity and lead to healthier dietary habits, smoking cessation and a higher quality of life.

It is unique that Central Denmark Region has assigned phase II CR as a local healthcare services. Thus, it is crucial to know more about performance in local healthcare services CR and whether all patients receive high-quality evidence-based services regardless of where they live. To our knowledge, no studies have examined the association between performance in different health pedagogical strategies and outcomes. This association is important to investigate when dramatic organisational changes in settings of evidence based interventions is implemented, as well as in relation to helping people with heart disease return to an active and satisfying everyday life. This study is unique and may inform and affect the way CR is organised and performed on a national and an international level to improve quality of care.

ELIGIBILITY:
Inclusion criteria:

We include all adult patients ( >18 years old) discharged from hospital with in Central Denmark Region between September 1, 2018 and July 31, 2019. Ischaemic Heart Disease will be defined according to the International Classification of Diseases version 10 (ICD-10): DI210, DI210A, DI210B, DI211, DI211A, DI211B, DI213, DI214, DI219, DI248, DI249, DI240, DI209, DI251, DI251B, and DI251. In 2016, this population represented approx. 2,700 patients.

Exclusion criteria:

People survive cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Adherence | During a 12 week programme
  Adherence to CR, defined as percentage of total prescribed sessions.

SECONDARY OUTCOMES:
Health-related quality of life | 4 times during 12 months after engaging Cardia Rehabilitation
  Questionnaire; HearQol The HeartQol questionnaire assesses health-related quality of life; physical and emotional condition. The HeartQoL questionnaire was first described in the literature in 2012. It is a 14-item assessment and evaluation system specific to IHD that assesses the impact of cardiac intervention on patient-reported health-related quality of life. HeartQoL consists of two subscales, a 10-item physical subscale and a 4-item emotional subscale. Scores range from 0 to 3 with higher scores indicating a better health-related quality of life. The HeartQol questionnaire has been validated in Danish patients with heart valve surgery.
Anxiety and depression | 4 times during 12 months after engaging Cardia Rehabilitation
  Questionnaire; HADS Hospital Anxiety and Depression Scale assesses states of depression and anxiety in the setting of an hospital medical outpatient clinic and primary care population. The scale consist of 14 items - seven concerning anxiety and seven concerning depression An analysis of scores on the two subscales of a further sample, in the same clinical setting, showed that a score of 0 to 7 for either subscale could be regarded as being in the normal range, a score of 11 or higher indicating probable presence ('caseness') of the mood disorder and a score of 8 to 10 being just suggestive of the presence of the respective state. The Hospital Anxiety and Depression Scale is a valid and reliable instrument that has been used across the world in cardiac and non-cardiac populations.
Coping | 4 times during 12 months after engaging Cardia Rehabilitation
  Questionnaire; PAM The Patient Activation Measure assesses the patients' activation level in four elements; knowledge, skills, confidence and behaviours. The scale consists of 13-items. The Patient Activation Measure identifies four different levels of activation. The Patient Activation Measure is a valid and reliable instrument that has been used across the world in populations with chronic diseases. The Patient Activation Measure is translated and validated in Danish setting.
Return to work | 12 months after ended Cardiac Rehabilitation
  Sick leave and work disability are registered in the Danish Register for Evaluation of Marginalisation (DREAM). DREAM includes all Danish citizens who have received social benefits or any other public benefits since July 1991. Transfer benefits, which can be grouped into five categories: Benefits to otherwise self-supporting individuals, labor market-related benefits, temporary health-related benefits (sickness benefit and vocational rehabilitation benefit), permanent health-related benefits (partial and full disability pension), and benefits related to old age or early retirement. If no transfer income is registered for a specific week, the person is considered to be self-supporting or on short-term sick-leave (less than 2 weeks). In Denmark, a citizen in the workforce (employed as well as unemployed) is entitled to sickness absence compensation, and in case the employee receives normal salary during sick leave, the employer receives a municipal reimbursement.
Cost-effectiveness | When patients enter intervention CR or usual CR and again 12 months after ended CR
  EQ-5D assesses health related quality of life and practical for economic evaluation. Patients are asked to complete the questionnaire at baseline and 12 months after the completed CR. EQ-5D was first introduced in 1990 by the EuroQol Group. The EQ-5D has been extensively used to assess patient utility in trials of new treatments. The index-based score is generated by applying societal preference weights to the health state classification completed by the patient that consists of five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), each with three levels of response or severity (no problems, some problems, or extreme problems). The ability to convert self classification responses into a single index score makes the EQ-5D practical for clinical and economic evaluation.
Completion | At the end of a 12 week rehabilitation program
  Completion is final CR assessment and discharge to long term management from primary health service. This information is obtained from the Central Denmark Region Cardiac Rehabilitation Database - recorded: yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Gjørup Pedersen, PhD, Principal Investigator — Defactum, Central Denmark Region
Locations (1):
- Charlotte Gjørup Pedersen, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No